CLINICAL TRIAL: NCT00726778
Title: Admixture Mapping of Ethnic and Racial Insulin Complex Outcomes
Acronym: AMERICO
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Jose Fernandez, UAB
Other Study IDs: F040109007; R01DK067426 (NIH)
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: race/ethnicity; insulin senistivity; genetic admixture; type 2 diabetes; obesity; body composition; Insulin dynamics; Racial/ethnic differences
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Three 5-ml blood samples will be obtained from each subject and sent to the Laboratory Core of the General Clinical Research Center to establish EBV lymphoblastoid cell lines and for DNA extraction. EBV lines will be kept at UAB for future genetic analysis. Extracted DNA will be sent to Dr. Mark Shriver at the Pennsylvania State University for genotyping of the ancestry informative markers (AIMs).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A, Observational: Healthy European American, African American, and Hispanic American children aged 7-12

SUMMARY:
The main objective of this study is to investigate the effect of genetic and environmental parameters on racial/ethnic differences in aspects of insulin secretion and action. The genetic component will be modeled by estimating the degree of European genetic admixture (ADM) obtained from approximately 50 ancestry informative markers (AIMs). The environmental components will be modeled by measuring energy intake (food intake), energy expenditure (physical activity) and socioeconomic status.

ELIGIBILITY:
Inclusion Criteria:

* African American, European American, or Hispanic American, aged 7-12, healthy, weight is equal to or greater than 25 Kg

Exclusion Criteria:

* Type 1 or 2 diabetes, polycystic ovary disease, disturbances in glucose or lipid metabolism disturbances
* Use of medication known to affect body composition or physical activity, diagnosis of genetic disorders known to affect body composition or fat distribution
* Use of tobacco, alcohol consumption in excess of 400 g per week
* Menstruated for more than a year prior to the recruitment; OR
* A medical history that counter-indicates inclusion of the study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 120 African Americans, 120 European Americans and 120 Hispanic Americans (60 males and 60 females per group). To minimize the influence of puberty on SI and AIRg, recruitment will be limited to individuals between ages 7-12, a range that based on previous observations from our team, categorize children from Tanner stage 1 and 2.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2004-05; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To test the role of European genetic admixture on measures of insulin action and response in a multiethnic group of prepubertal children. | 5 years
To investigate whether the impact of energy intake, energy expenditure and socioeconomic status on proxy measures of insulin sensitivity and/or action differ as a function of European ADM in prepubertal children | 5 years
To test phenotype-genotype associations between each one of the AIMs and measures of FI, SI and AIRg after adjusting for body composition in a sample of AA, HA and EA prepubertal children. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jose Fernandez, Ph.D., Principal Investigator — UA B
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Cardel M, Lemas DJ, Jackson KH, Friedman JE, Fernandez JR. Higher Intake of PUFAs Is Associated with Lower Total and Visceral Adiposity and Higher Lean Mass in a Racially Diverse Sample of Children. J Nutr. 2015 Sep;145(9):2146-52. doi: 10.3945/jn.115.212365. Epub 2015 Aug 12. PMID 26269238
- [Derived] Kell KP, Cardel MI, Bohan Brown MM, Fernandez JR. Added sugars in the diet are positively associated with diastolic blood pressure and triglycerides in children. Am J Clin Nutr. 2014 Jul;100(1):46-52. doi: 10.3945/ajcn.113.076505. Epub 2014 Apr 9. PMID 24717340